CLINICAL TRIAL: NCT05587569
Title: Radiographic and Patient Reported Outcomes Following Combined Adductoplasty™ and Lapiplasty® Procedures for Correction of Metatarsus Adductus and Hallux Valgus (MTA3D)
Brief Title: Outcomes Following Combined Adductoplasty™ and Lapiplasty® (MTA3D)
Acronym: MTA3D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Treace Medical Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2022-1
Record Dates: First submitted 2022-10-10; First posted 2022-10-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Metatarsus Adductus; Hallux Valgus
Keywords: Metatarsus Adductus; Hallux Valgus; MTA3D
MeSH Terms: conditions — Metatarsus Varus; Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Treatment of metatarsus adductus and hallux valgus with the Adductoplasty™ Procedure in combination with the Lapiplasty® Procedure — Patients 14 years of age or older with symptomatic metatarsus adductus and hallux valgus will be eligible to participate based on the inclusion/exclusion criteria established in the study protocol. Anticipated study duration will be 5 years post index procedure.
  Other Names: Adductoplasty™ Procedure in combination with the Lapiplasty® Procedure

SUMMARY:
Prospective, multicenter, unblinded study to evaluate outcomes of the Adductoplasty™ Procedure in combination with the Lapiplasty® Procedure for patients in need of metatarsus adductus and hallux valgus correction.

Up to 80 subjects will be treated in this study at up to 13 clinical sites. Patients 14 years of age or older with symptomatic metatarsus adductus and hallux valgus will be eligible to participate based on the inclusion and exclusion criteria defined in the study protocol.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate outcomes of the Adductoplasty™ Procedure combined with the Lapiplasty® Procedure for patients in need of hallux valgus and metatarsus adductus surgery:

1. To evaluate the quality of life and pain scores following the Adductoplasty™ Procedure in combination with the Lapiplasty® Procedure.
2. To determine whether the Adductoplasty™ Procedure in combination with the Lapiplasty® Procedure, effectively corrects and maintains triplane anatomical alignment of the 1st, 2nd and 3rd metatarsals, the hallux position, the sesamoid position, and the foot width.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females ≥14 years old at the time of consent
2. Closed physeal plates at the time of consent
3. Intermetatarsal angle is ≥8.0˚; OR True IMA of >10°, (IMA+MTA-15=True IMA)
4. Hallux valgus angle is ≥12.0˚
5. Metatarsus adductus angle based on Sgarlatos method ≥15°
6. Willing and able to adhere to post-op care instructions
7. Capable of completing self-administered questionnaires
8. Acceptable surgical candidate, including use of general anesthesia
9. Female patients must be of non-childbearing potential or have a negative pregnancy test in accordance with hospital standards prior to the Index Procedure
10. Willing and able to schedule index procedure within 3 months of consent and able to return for scheduled follow-up visits
11. Willing and able to provide written informed consent
12. Patient agrees to refrain from any reconstructive procedures on contralateral foot for minimum of 6 months post index procedure

Exclusion Criteria:

1. Previous surgery for hallux valgus on operative side
2. Previous surgeries on operative foot involving fusion of foot or ankle joints (other than hammertoe, lesser toes/digits, or posterior muscle lengthening)
3. Moderate-severe osteoarthritis of the foot or ankle outside of the 1st, 2nd or 3rd tarsometatarsal joints
4. Severe osteoarthritis of the 1st, 2nd or 3rd tarsometatarsal joints
5. Any deformity of the hindfoot or midfoot that represents a pathological condition that may affect the outcome of the tarsometatarsal realignment, or a condition that requires concomitant surgical correction
6. BMI >40 kg/m²
7. Current nicotine user in any form including vaping, smoking, oral ingestion or use of nicotine patch
8. Current clinical diagnosis of diabetes or currently taking medication for treatment of diabetes
9. Current clinical diagnosis of peripheral neuropathy
10. Current clinical diagnosis of fibromyalgia
11. Current clinical diagnosis of Complex Regional Pain Syndrome/Reflex Sympathetic Dystrophy (CRPS/RSD)
12. Current uncontrolled hypothyroidism
13. Current clinical diagnosis of chronic dependent edema
14. Previously sensitized to titanium
15. Currently taking oral steroids or rheumatoid biologics
16. Currently taking immunosuppressant drugs
17. Insufficient quantity or quality of bone to permit stabilization, conditions that inhibit healing (not including pathological fractures) and conditions causing poor blood supply such as peripheral vascular disease
18. Active, suspected, or latent infection in the affected area
19. Use of synthetic or allogenic bone graft substitutes
20. Use of non-Treace products for Index Procedure
21. Additional bone procedure needed during the index procedure to complete correction [first MTP fusion, calcaneal osteotomy, traditional medial eminence resection, additional metatarsal or tarsal bone osteotomy or fusion (other than Weil osteotomies)];
22. Scheduled to undergo a same-day bilateral procedure
23. Patient has previously been enrolled into this study for a contralateral procedure
24. Scheduled for any concomitant procedure that would alter patient's ability to weight-bear post-procedure
25. Patient is actively involved with a workman's compensation case or is currently involved in litigation
26. Patient is currently in, or has participated in, a clinical study in the last 30 days prior to signing informed consent or is considering participation in another research protocol during this study. Exceptions to this include survey clinical studies with no treatment or if subject is greater than 12 months post procedure in either the Treace ALIGN3D™ or Mini3D™ Study without ongoing protocol defined AE
27. Patient has a condition or finding that, in the opinion of the Investigator, may jeopardize the patient's well-being, the soundness of this clinical study, or could interfere with provision of informed consent, completion of tests, therapy, or follow-up

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic recurrence of hallux valgus deformity with metatarsus adductus will be evaluated at 24 months for subjects wtih successful correction | 24 Months
  Successful correction is defined as two of the following three criteria: measured IMA <9.0°, HVA <15.0°, and TSP as ≤3 at 6 months post Adductoplasty® Procedure and Lapiplasty® Procedure. Recurrence at 24 months is defined by HVA >15.0°.

SECONDARY OUTCOMES:
Radiographic Recurrence | 24 Months
  Radiographic recurrence of hallux valgus deformity at 24 months defined by HVA >20°.
Union vs non-Union | 12 Months
  Evaluate clinical/radiographic healing (union vs non-union). Non-union is defined as pain and lucency at the 1st, 2nd, and/or 3rd TMT joint at 12 months post- Adductoplasty® Procedure and Lapiplasty® Procedure.
Clinical Complications | 60 Months
  Clinical complications due to system implants the post-op instructions or health conditions that could affect other outcome measures.
Weight-Bearing Recovery Time | 12 Months
  Assessment of weight-bearing recovery time following the procedures. Weight-bearing will be measured in days and recorded based upon individual surgeon recovery protocol.
Time to Weight-Bear in Boot | 6 Weeks
  Time to start of weight-bearing in boot, in days.
Time to Weight-Bear in Shoes | 8 Weeks
  Time to start of weight-bearing in shoes, in days.
Time to Return to Unrestricted Activity | 6 weeks - 6 months, post Lapiplasty® Procedure
  Time to return to full unrestricted activity, in days.
Change in Pain | 0-3 weeks, 6 weeks, 4 months, 6 months, 12 months, 24 months, 36 months, 48 months and 60 months post- Adductoplasty™ Procedure in combination with the Lapiplasty® Procedure, in comparison to baseline visit pain.
  Change in pain at the base of the big toe (bunion related), as well as the midfoot region for the operative foot only, assessed via the Visual Analog Scale (VAS) with 0-10 minimum and maximum values - with 0 being a better outcome and 10 being a worse outcome.
Change in Quality of Life | 6 months, 12 months, 24 months, 36 months, 48 months and 60 months post-Adductoplasty™ Procedure and Lapiplasty® Procedure, in comparison to baseline visit
  Change in Quality of Life, (PROMIS-29/PROMIS-25 and MOxFQ) defined as the total domain score measured.
Change in Range of Motion | 12 months, 24 months, 36 months, 48 months and 60 months post- Adductoplasty™ Procedure and Lapiplasty® Procedure, in comparison to baseline visit
  Change in Range of Motion - 1st MTP dorsiflexion and plantarflexion
Change in Osseous Foot Width | 12 months and 24 months post - Adductoplasty™ Procedure and Lapiplasty® Procedure, in comparison to baseline visit
  Change in osseous foot width - radiographically

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dayton, DPM, Principal Investigator — Foot and Ankle Center of Iowa; Mark Easley, MD, Principal Investigator — Duke University
Locations (9):
- United States (9):
  - Foot and Ankle Center of the Rockies, Greeley, Colorado
  - Foot and Ankle Center of Iowa, Ankeny, Iowa
  - Coastal Maine Foot and Ankle, Yarmouth, Maine
  - JCMG - Jefferson City Medical Group, Jefferson City, Missouri
  - Duke Orthopaedics Arringdon, Morrisville, North Carolina
  - Ohio Foot and Ankle Center, Canton, Ohio
  - Ohio Foot and Ankle Center, Stow, Ohio
  - Greater Pittsburgh Foot and Ankle Center, Wexford, Pennsylvania
  - Foot and Ankle Associates of North Texas - Keller, Keller, Texas

IPD SHARING:
Plan to Share IPD: No